CLINICAL TRIAL: NCT00498550
Title: Cannabis and Schizophrenia: Effects of Clozapine
Brief Title: Treatment of Schizophrenia and Comorbid Cannabis Use Disorder: Comparing Clozapine to Treatment-as-Usual
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Missouri, Kansas City (Other); VA Medical Center-West Los Angeles (U.S. Federal Agency); University of South Carolina (Other)
Responsible Party: Principal Investigator, Alan Green, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCT00149955; R01DA013196 (NIH); DPMCDA; NCT00149955 (obsolete NCT alias)
Record Dates: First submitted 2007-07-06; First posted 2007-07-10 (Estimated); Results first posted 2012-01-19 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Schizophrenia; Dual Diagnosis; Schizoaffective Disorder; Psychotic Disorder; Cannabis Abuse
Keywords: Clozapine; Schizophrenia; Dual Diagnosis; Substance Abuse; Cannabis Abuse
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Marijuana Abuse; Substance-Related Disorders | interventions — Clozapine; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clozapine (Experimental): Clozapine, Clozaril
  Interventions: Drug: Clozapine
- Treatment as usual (Active Comparator): Treatment as usual with any antipsychotic other than Clozapine.
  Interventions: Drug: Treatment as usual

INTERVENTIONS:
Drug: Clozapine — Clozapine up to 550mg per day
  Other Names: Clozaril
  Arms: Clozapine
Drug: Treatment as usual — Remain on pre-study antipsychotic treatment
  Arms: Treatment as usual

SUMMARY:
Many individuals with schizophrenia also suffer from marijuana addiction. Clozapine, an atypical antipsychotic medication, may prove useful at preventing drug relapse in schizophrenic individuals who are seeking treatment for marijuana addiction. The purpose of this study is to compare the effectiveness of clozapine, vs. treatment-as-usual with other oral antipsychotics at reducing marijuana use in schizophrenic individuals.

DETAILED DESCRIPTION:
Individuals with schizophrenia have a high risk of becoming addicted to drugs; between 13 to 42% of schizophrenics are addicted to marijuana. These individuals often have difficulties adhering to a substance abuse treatment program, and have an increased chance of marijuana relapse. Marijuana use by schizophrenics has also been associated with clinical exacerbations, noncompliance with antipsychotic medications, poor global functioning, and increased rehospitalization rates. While antipsychotic medications are often effective in controlling symptoms of schizophrenia, they are not always effective in preventing substance abuse. Clozapine, an atypical antipsychotic drug, is currently used to treat schizophrenia. Preliminary research has shown that clozapine is more successful at reducing drug relapse rates in individuals with schizophrenia, as compared to other antipsychotic medications, including olanzapine and risperidone. The purpose of this study is to compare the effectiveness of clozapine as compared to other oral antipsychotic treatment, including combinations of up to two antipsychotics, in reducing marijuana use in schizophrenic individuals.

This study will enroll individuals with schizophrenia who are currently taking any oral antipsychotic other than clozapine, including those taking up to two oral antipsychotic, and who are also addicted to marijuana. The study will begin with a 1-week assessment phase, during which all participants will continue taking olanzapine or risperidone. Participants will undergo a physical examination and have blood drawn for laboratory tests. Information pertaining to their medical, psychiatric, and substance use history will also be collected. Urine tests and breathalyzers will be used to screen for the presence of alcohol and drugs. Following the assessment phase, participants will be randomly assigned to switch to clozapine or remain on their prestudy antipsychotic for 12 weeks. Participants remaining on their prestudy antipsychotic treatment will continue to receive the same dose for the entire study. Participants taking clozapine will initially receive a daily dose of 12.5 mg, which will be increased to a maximum of 400 mg per day, as tolerated. Study visits will take place once a week. At each visit, medication side effects, physical and psychological symptoms, substance use, treatment services received, and living situation will be assessed. Blood will be drawn for laboratory tests. Drug and alcohol levels will be monitored three times a week through urine and breathalyzer tests. Quality of life questionnaires will be administered once a month.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statical Manual of Mental Disorders IV (DSM-IV) diagnostic criteria for schizophrenia or schizoaffective disorder
* Meets diagnostic criteria for marijuana use disorder, as determined by a rating of 3 or higher on the Drug Use Scale (Abuse or Dependence)
* Used marijuana on 5 or more days during the 3 weeks prior to study entry
* Taking any oral antipsychotic other than clozapine in the month prior to study entry. (Patients may take a second oral antipsychotic medication, if approved by the Medication Adjustment Group)
* If female, willing to use effective contraception throughout the study

Exclusion Criteria:

* Unable to take clozapine for medical reasons, including previous clozapine-induced granulocytopenia, myeloproliferative disorder, white blood cell count less than 3500/mm3, or history of seizures
* Currently taking clozapine
* Currently taking other psychotropic medications for the treatment of substance use (e.g., disulfiram, naltrexone, acamprosate, inderol, tegretol, topiramate, and pramipexole)
* Participated in a clinical trial of an investigational drug within 30 days of study entry
* Currently participating in a psychosocial intervention clinical trial
* Has medical or legal problems that may entail a jail or hospital stay during the study
* Has a developmental disability that would make study participation difficult
* Currently enrolled in a live-in treatment program for substance use disorders
* Pregnant or plans to become pregnant during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2000-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Green, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (4):
- United States (4):
  - West LA VAHCS, Los Angeles, California
  - University Missouri, Kansas City, Missouri
  - Mental Health Center of Greater Manchester, Manchester, New Hampshire
  - University South Carolina, Columbia, South Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clozapine | Treatment as Usual
Started | 15 | 16
Completed | 15 (13 of 15 received clozapine all 12 visits, two discontinued clozapine early but remained in study.) | 15
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clozapine | Treatment as Usual | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (10.0) | 39.0 (10.2) | 36 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 12 | 12 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Average Over Time of Intensity of Cannabis Use (Used to Evaluate Treatment Efficacy)
Description: Intensity of cannabis use is obtained for each week retrospectively as the number of joints smoked during the prior week (assessed by the Timeline Followback Scale). Mixed models are used to obtain estimates of efficacy from the partial data provided by each subject while adherent to assigned treatment (under the 'missing at random' assumption). The 'explanatory' estimands (target of the mixed model estimation) are defined in terms of population quantities that would have occurred had all subjects remained on assigned treatment throughout the study. The point estimate for each arm is reported under Number.
Time Frame: Week 1 to week 12
Measure: Number (95% Confidence Interval); unit: Joints per week
Arm/Group | Clozapine | Treatment as Usual
Number analyzed (Participants) | 15 | 16
Joints per week | 0.02 [-2.1 to 2.5] | 4.56 [-0.2 to 9.3]
Statistical Analysis 1: Comparison: Clozapine vs Treatment as Usual; Test type: Superiority; p = .088, Mixed Models Analysis; difference in treatment means = -4.54, Standard Error of Mean 2.57 — We report the estimated coefficient for difference in treatment means in a mixed model and its standard error

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Clozapine | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 4/15 | 4/16
Other Adverse Events (participants affected / at risk) | 15/15 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clozapine (N=15) | Treatment as Usual (N=16)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Psychiatric Disorder - Other: Accidental Overdose (Psychiatric disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 1 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clozapine (N=15) | Treatment as Usual (N=16)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 5 (8) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 2 (3) | 2 (2)
Fatigue (General disorders) | 3 (3) | 0 (0)
Flu Like Symptoms (General disorders) | 0 (0) | 2 (2)
Gastrointestinal Disorder - Other: Hypersalivation (Gastrointestinal disorders) | 10 (11) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Irritability (General disorders) | 1 (1) | 1 (1)
Libido Decreased (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Musculoskeletal And Connective Tissue Disorder - Other: Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (5) | 1 (1)
Nervous Sytem Disorder - Other: Unusual Dream Activity (Nervous system disorders) | 0 (0) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 9 (12) | 2 (2)
Urinary Incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Weight Gain (Investigations) | 6 (7) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No